CLINICAL TRIAL: NCT04910074
Title: LLLT Effects on Inferior Alveolar Nerve (IAN) Recovery Post-orthognathic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI terminated study due to lack of resources.
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-12990
Record Dates: First submitted 2021-05-28; First posted 2021-06-02 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Mandible; Deformity; Surgical Healing; Orthognathic Surgery; Nerve Injury
Keywords: orthognathic; lllt
MeSH Terms: conditions — Congenital Abnormalities | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: intervention vs placebo
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcomes assessor will be blinded to which group participants belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Low-level therapy intervention (Experimental): Patients will receive low-level laser therapy on the skin overlying the mandible for 40 seconds per side. All other post-operative care will be as per clinic routine.
  Interventions: Device: Low-level laser therapy
- dummy intervention (Placebo Comparator): Patients will receive no dose of laser, but the handpiece will be used against their skin top mimic the LLLT. All other post-operative care will be as per clinic routine.
  Interventions: Device: Dummy LLLT

INTERVENTIONS:
Device: Low-level laser therapy — The proposed LLLT protocol will use the Biolase Epic X, an InGaAsP diode laser (940nm) using the pain relief handpiece, a device which has received FDA approval (GUDID 00647529002537) for the treatment of pain, muscle relaxation and healing via increased local circulation. The LLLT will be administered to the experimental group at 30 j/cm2. The laser will be applied extraorally, on the skin overlying the mandible. Application will be for 40 seconds per side, with 10 seconds administered in four places along the jawline, 1 cm apart starting from the gonial angle.
  Arms: Low-level therapy intervention
Device: Dummy LLLT — The Biolase Epic X with pain relief handpiece will be applied with no power extraorally, on the skin overlying the mandible. Application will be for 40 seconds per side, with 10 seconds administered in four places along the jawline, 1 cm apart starting from the gonial angle.
  Arms: dummy intervention

SUMMARY:
Low-level laser therapy (LLLT) is a well-studied technique that has been shown to improve recovery time and reduce pain and swelling in patients undergoing surgery, including orthognathic surgery, and has no known negative effects. This study will use two groups with patients randomly assigned to either the study group, receiving LLLT, or one receiving a placebo treatment, after they have lower jaw surgery. Measurements will be taken at 24 hours, 1 week, 2 week, 3 week, 4 week, 5 week, and 6 week post-op exams to check pain, swelling and nerve function, and the two groups will be compared to see if the LLLT group has any difference

DETAILED DESCRIPTION:
Low-level laser therapy (LLLT) is a well-studied technique to induce biomodulation of pain and wound healing. The technique has been shown to improve recovery time and reduce pain and swelling in patients undergoing surgery, including orthognathic surgery, and has no known negative effects. Previous studies have used split-mouth designs, short follow-up periods or, often, both. This study aims to have two groups, one receiving LLLT and one receiving a dummy treatment, at 24 hours, 1 week, 2 week, 3 week, 4 week, 5 week, and 6 week post-op exams. At each visit, pain (via VAS), swelling (measured from the midpoint of the chin to the base of the ear, bilaterally), and nerve function (using a soft and hard sensory test, in 8 regions of the mandible and lower lip) will be performed, with additional measurements at 8 weeks and 20 weeks. The measurements will be analyzed for statistical differences between the LLLT intervention group and non-intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mandibular surgery with bilateral sagittal split osteotomies

Exclusion Criteria:

* patients must be free from pre-operative inferior alveolar neurosensory deficiencies
* intra-operative accidental fracture or rupture of the inferior alveolar nerve

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Levine, DMD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, Department of Dentistry and Oral Surgery, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Agostino A, Trevisiol L, Gugole F, Bondi V, Nocini PF. Complications of orthognathic surgery: the inferior alveolar nerve. J Craniofac Surg. 2010 Jul;21(4):1189-95. doi: 10.1097/SCS.0b013e3181e1b5ff. PMID 20613608
- [Background] Haghighat A, Khosrawi S, Tamizifar A, Haghighat M. RETRACTED: Does Low-Level Laser Photobiomodulation Improve Neurosensory Recovery After Orthognathic Surgery? A Clinical Trial With Blink Reflex. J Oral Maxillofac Surg. 2021 Mar;79(3):685-693. doi: 10.1016/j.joms.2020.11.025. Epub 2020 Nov 30. PMID 33358708 (Retraction: PMID 34862008 J Oral Maxillofac Surg. 2021 Dec;79(12):2606)
- [Background] Gasperini G, Rodrigues de Siqueira IC, Rezende Costa L. Does low-level laser therapy decrease swelling and pain resulting from orthognathic surgery? Int J Oral Maxillofac Surg. 2014 Jul;43(7):868-73. doi: 10.1016/j.ijom.2014.02.015. Epub 2014 Mar 25. PMID 24679851
- [Background] Khullar SM, Emami B, Westermark A, Haanaes HR. Effect of low-level laser treatment on neurosensory deficits subsequent to sagittal split ramus osteotomy. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Aug;82(2):132-8. doi: 10.1016/s1079-2104(96)80215-0. PMID 8863301
- [Background] Firoozi P, Keyhan SO, Kim SG, Fallahi HR. Effectiveness of low-level laser therapy on recovery from neurosensory disturbance after sagittal split ramus osteotomy: a systematic review and meta-analysis. Maxillofac Plast Reconstr Surg. 2020 Dec 17;42(1):41. doi: 10.1186/s40902-020-00285-0. PMID 33331972
- [Background] Ezzati K, Fekrazad R, Raoufi Z. The Effects of Photobiomodulation Therapy on Post-Surgical Pain. J Lasers Med Sci. 2019 Spring;10(2):79-85. doi: 10.15171/jlms.2019.13. Epub 2019 Feb 25. PMID 31360374
- [Background] Ozen T, Orhan K, Gorur I, Ozturk A. Efficacy of low level laser therapy on neurosensory recovery after injury to the inferior alveolar nerve. Head Face Med. 2006 Feb 15;2:3. doi: 10.1186/1746-160X-2-3. PMID 16480503
- [Background] Esteves Pinto Faria P, Temprano A, Piva F, Sant'ana E, Pimenta D. Low-level laser therapy for neurosensory recovery after sagittal ramus osteotomy. Minerva Stomatol. 2020 Jun;69(3):141-147. doi: 10.23736/S0026-4970.20.04289-2. Epub 2020 Mar 16. PMID 32181610
- [Background] Bittencourt MA, Paranhos LR, Martins-Filho PR. Low-level laser therapy for treatment of neurosensory disorders after orthognathic surgery: A systematic review of randomized clinical trials. Med Oral Patol Oral Cir Bucal. 2017 Nov 1;22(6):780-787. doi: 10.4317/medoral.21968. PMID 29053658
- [Background] Hamid MA. Low-level Laser Therapy on Postoperative Pain after Mandibular Third Molar Surgery. Ann Maxillofac Surg. 2017 Jul-Dec;7(2):207-216. doi: 10.4103/ams.ams_5_17. PMID 29264287
- [Background] Boutault F, Diallo R, Marecaux C, Modiga O, Paoli JR, Lauwers F. [Neurosensory disorders and functional impairment after bilateral sagittal split osteotomy: role of the anatomical situation of the alveolar pedicle in 76 patients]. Rev Stomatol Chir Maxillofac. 2007 Jun;108(3):175-82; discussion 182. doi: 10.1016/j.stomax.2006.11.006. Epub 2007 Apr 19. French. PMID 17448510
- [Background] Al-Bishri A, Barghash Z, Rosenquist J, Sunzel B. Neurosensory disturbance after sagittal split and intraoral vertical ramus osteotomy: as reported in questionnaires and patients' records. Int J Oral Maxillofac Surg. 2005 May;34(3):247-51. doi: 10.1016/j.ijom.2004.06.009. PMID 15741031
- [Background] Al-Bishri A, Rosenquist J, Sunzel B. On neurosensory disturbance after sagittal split osteotomy. J Oral Maxillofac Surg. 2004 Dec;62(12):1472-6. doi: 10.1016/j.joms.2004.04.021. PMID 15573346
- [Background] Reddy GK. Photobiological basis and clinical role of low-intensity lasers in biology and medicine. J Clin Laser Med Surg. 2004 Apr;22(2):141-50. doi: 10.1089/104454704774076208. PMID 15165389
- [Background] Kuroyanagi N, Miyachi H, Ochiai S, Kamiya N, Kanazawa T, Nagao T, Shimozato K. Prediction of neurosensory alterations after sagittal split ramus osteotomy. Int J Oral Maxillofac Surg. 2013 Jul;42(7):814-22. doi: 10.1016/j.ijom.2012.11.016. Epub 2012 Dec 21. PMID 23265759
- [Background] Baas EM, Horsthuis RB, de Lange J. Subjective alveolar nerve function after bilateral sagittal split osteotomy or distraction osteogenesis of mandible. J Oral Maxillofac Surg. 2012 Apr;70(4):910-8. doi: 10.1016/j.joms.2011.02.107. Epub 2011 Jul 16. PMID 21763047
- [Background] TRAUNER R, OBWEGESER H. The surgical correction of mandibular prognathism and retrognathia with consideration of genioplasty. II. Operating methods for microgenia and distoclusion. Oral Surg Oral Med Oral Pathol. 1957 Aug;10(8):787-92; contd. No abstract available. PMID 13452398

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-level Therapy Intervention: Patients will receive low-level laser therapy on the skin overlying the mandible for 40 seconds per side. All other post-operative care will be as per clinic routine.
  Low-level laser therapy (LLLT): The proposed LLLT protocol will use the Biolase Epic X, an InGaAsP diode laser (940nm) using the pain relief handpiece, a device which has received FDA approval (GUDID 00647529002537) for the treatment of pain, muscle relaxation and healing via increased local circulation. The LLLT will be administered to the experimental group at 30 j/cm2. The laser will be applied extraorally, on the skin overlying the mandible. Application will be for 40 seconds per side, with 10 seconds administered in four places along the jawline, 1 cm apart starting from the gonial angle.
- Sham Intervention: Patients will receive no dose of laser, but the handpiece will be used against their skin top mimic the LLLT. All other post-operative care will be as per clinic routine.
  Sham LLLT: The Biolase Epic X with pain relief handpiece will be applied with no power extraorally, on the skin overlying the mandible. Application will be for 40 seconds per side, with 10 seconds administered in four places along the jawline, 1 cm apart starting from the gonial angle.
Period: Overall Study
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Started | 12 | 13
Completed | 0 | 0
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-level Therapy Intervention | Sham Intervention | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25
Inferior Alveolar Nerve (IAN) Function for Soft Stimuli [Count of Participants; unit: Participants] — IAN function for soft stimuli was assessed by brushing a cotton swab along a 2cm path of the skin of the mandible and lower lip in 8 regions along the lower jaw. Regions right and left 1, 2 and 3 are on the skin of lower face, 1 cm apart, starting on the midline, and right and left region 4 is the lower lip, separated at the midline. Right and left regions were identified as R1, R2, R3, R4 and L1, L2, L3, and L4, respectively. Patients responded as to whether they were able to feel the cotton swab using a binary Yes(+) or No(-) response. The number of patients who responded Yes is summarized. Population: Swab samples were only collected from 10 patients in the Sham intervention arm with the exception of region L2 and region L3 samples which were only collected from 9 patients in the Sham intervention arm.
  Participants
    R1: number analyzed (Participants) | 12 | 10 | 22
    R1 | 12 | 10 | 22
    R2: number analyzed (Participants) | 12 | 10 | 22
    R2 | 12 | 10 | 22
    R3: number analyzed (Participants) | 12 | 10 | 22
    R3 | 12 | 10 | 22
    R4: number analyzed (Participants) | 12 | 10 | 22
    R4 | 12 | 10 | 22
    L1: number analyzed (Participants) | 12 | 10 | 22
    L1 | 12 | 10 | 22
    L2: number analyzed (Participants) | 12 | 9 | 21
    L2 | 12 | 9 | 21
    L3: number analyzed (Participants) | 12 | 9 | 21
    L3 | 12 | 9 | 21
    L4: number analyzed (Participants) | 12 | 10 | 22
    L4 | 12 | 10 | 22
Inferior Alveolar Nerve (IAN) Function for Hard Stimuli [Count of Participants; unit: Participants] — IAN function for hard stimuli was assessed by pressing a toothpick into the skin of the mandible and lower lip in 8 regions along the lower jaw. Regions right and left 1, 2, and 3 are on the skin of the lower face, 1 cm apart, starting on the midline, and right and left region 4 is the lower lip, separated at the midline. Right and left regions were abbreviated as R1, R2, R3, R4 and L1, L2, L3, and L4, respectively. Patients responded as to whether they were able to feel the toothpick using a binary Yes (+) or No (-) response. The number of patients who responded Yes (+) is summarized. Population: Toothpick samples were collected from all 12 patients in the Low-level therapy intervention arm with the exception of a region L4 sample in one patient. Toothpick samples were only collected from 10 patients in the Sham intervention arm.
  Participants
    R1: number analyzed (Participants) | 12 | 10 | 22
    R1 | 12 | 10 | 22
    R2: number analyzed (Participants) | 12 | 10 | 22
    R2 | 12 | 10 | 22
    R3: number analyzed (Participants) | 12 | 10 | 22
    R3 | 12 | 10 | 22
    R4: number analyzed (Participants) | 12 | 10 | 22
    R4 | 12 | 10 | 22
    L1: number analyzed (Participants) | 12 | 10 | 22
    L1 | 12 | 10 | 22
    L2: number analyzed (Participants) | 12 | 10 | 22
    L2 | 12 | 10 | 22
    L3: number analyzed (Participants) | 12 | 10 | 22
    L3 | 12 | 10 | 22
    L4: number analyzed (Participants) | 11 | 10 | 21
    L4 | 11 | 10 | 21
Pre-Operative Pain [Mean (Standard Deviation); unit: score on a scale] — Pre-operative pain at baseline was reported via a Visual Analog Scale (VAS) response on the questionnaire. Using the VAS, patients rated the intensity of the pain on each side of the mandible (right and left). Possible VAS scores ranged from 0 (complete absence of pain) to 10 (maximum amount of pain imaginable). Results were summarized by study arm using basic descriptive statistics. Population: Pain intensity data at baseline was only able to be collected from 5 patients in the Low-level therapy intervention arm and 9 patients in the Sham intervention arm.
  score on a scale
    Right Side: number analyzed (Participants) | 5 | 9 | 14
    Right Side | 0.4 (0.5) | 0.1 (0.3) | 0.2 (0.4)
    Left Side: number analyzed (Participants) | 5 | 9 | 14
    Left Side | 0.4 (0.5) | 0.1 (0.3) | 0.2 (0.4)
Pre-Operative Mandibular Swelling [Mean (Standard Deviation); unit: millimeters] — Pre-operative mandibular swelling was measured using soft measuring tape. The extent of pre-operative swelling at baseline was measured from the tip of the chin to the base of the earlobe bilaterally (right and left). Measurements were recorded in millimeters (mm) and results summarized by study arm using basic descriptive statistics. Population: Pre-operative mandibular swelling was able to be assessed in 6 of 12 patients in the Low-level therapy intervention arm and 8 of 13 patients in the Sham intervention arm.
  millimeters
    Right Side: number analyzed (Participants) | 6 | 8 | 14
    Right Side | 149 (9.91) | 158 (14.2) | 153 (12.3)
    Left Side: number analyzed (Participants) | 6 | 8 | 14
    Left Side | 151 (9.13) | 160 (15.6) | 155 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: IAN function for soft stimuli was assessed by brushing a cotton swab along a 2cm path of the skin of the mandible and lower lip in 8 regions along the lower jaw. Regions right and left 1, 2 and 3 are on the skin of lower face, 1 cm apart, starting on the midline, and right and left region 4 is the lower lip, separated at the midline. Right and left regions were identified as R1, R2, R3, R4 and L1, L2, L3, and L4, respectively. Patients responded as to whether they were able to feel the cotton swab using a binary Yes (+) or No (-) response. The number of patients who responded Yes is summarized by study arm.
Time Frame: 24 hours post-surgery
Population: 24-hour post-surgical follow-up visits were not conducted during this study. Many patients were still admitted at 24 hours post-procedure and were unable to be brought into the dental clinic. In addition, the instruments and equipment required to conduct this assessment were not available in the hospital in-patient rooms. As a result, cotton swab samples were not obtained from any of the patients at 24 hours post-surgery and there is no IAN function for soft stimuli results data to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 1 week post-surgery
Population: Swab samples were able to be collected from regions R1, R4, L1, and L4 in all 12 patients and from regions R2, R3, L2, and L3 in 11 of 12 patients in the Low-level therapy intervention arm who attended their Week 1 visit. Swab samples were able to be collected from regions R2, R3, L2, and L3 in all 8 patients and from regions R1, R4, L1, and L4 in 7 of 8 patients in the Sham intervention arm who attended their Week 1 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 12 | 8
Participants
  R1: number analyzed (Participants) | 12 | 7
  R1 | 10 | 3
  R2: number analyzed (Participants) | 11 | 8
  R2 | 11 | 8
  R3: number analyzed (Participants) | 11 | 8
  R3 | 11 | 6
  R4: number analyzed (Participants) | 12 | 7
  R4 | 7 | 2
  L1: number analyzed (Participants) | 12 | 7
  L1 | 8 | 1
  L2: number analyzed (Participants) | 11 | 8
  L2 | 11 | 8
  L3: number analyzed (Participants) | 11 | 8
  L3 | 11 | 8
  L4: number analyzed (Participants) | 12 | 7
  L4 | 8 | 2

3. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 2 weeks post-surgery
Population: Swab samples were able to be collected from all regions in all 10 patients in the Low-level therapy intervention arm who attended their Week 2 visit. Swab samples were able to be collected from all regions in all 9 patients in the Sham intervention arm with the exception of regions R4 and L4 in which swab samples were able to be collected from 8 of 9 patients who attended their Week 2 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 10 | 9
Participants
  R1 | 8 | 6
  R2 | 9 | 9
  R3 | 10 | 9
  R4: number analyzed (Participants) | 10 | 8
  R4 | 7 | 5
  L1 | 7 | 4
  L2 | 10 | 9
  L3 | 10 | 9
  L4: number analyzed (Participants) | 10 | 8
  L4 | 6 | 3

4. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 3 weeks post-surgery
Population: Swab samples were able to be collected from all regions in all 10 patients in the Low-level therapy intervention arm and from all regions in all 8 patients in the Sham intervention arm who attended their Week 3 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 10 | 8
Participants
  R1 | 7 | 5
  R2 | 10 | 8
  R3 | 10 | 8
  R4 | 8 | 6
  L1 | 7 | 3
  L2 | 10 | 7
  L3 | 10 | 7
  L4 | 7 | 4

5. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 4 weeks post-surgery
Population: Swab samples were able to be collected from all regions in all 8 patients in the Low-level therapy intervention arm and from all regions in all 9 patients in the Sham intervention arm who attended their Week 4 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 8 | 9
Participants
  R1 | 5 | 6
  R2 | 8 | 9
  R3 | 8 | 9
  R4 | 7 | 7
  L1 | 4 | 6
  L2 | 8 | 9
  L3 | 8 | 9
  L4 | 5 | 5

6. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 5 weeks post-surgery
Population: Swab samples were able to be collected from regions L1 and L4 in all 7 patients and from regions R1, R2, R3, R4, L2, and L3 in 6 of 7 patients in the Low-level therapy intervention arm who attended their Week 5 visit. Swab samples were able to be collected from all regions in all 6 patients in the Sham intervention arm who attended their Week 5 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 7 | 6
Participants
  R1: number analyzed (Participants) | 6 | 6
  R1 | 6 | 3
  R2: number analyzed (Participants) | 6 | 6
  R2 | 6 | 6
  R3: number analyzed (Participants) | 6 | 6
  R3 | 6 | 6
  R4: number analyzed (Participants) | 6 | 6
  R4 | 6 | 4
  L1 | 3 | 4
  L2: number analyzed (Participants) | 6 | 6
  L2 | 6 | 6
  L3: number analyzed (Participants) | 6 | 6
  L3 | 6 | 6
  L4 | 3 | 4

7. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 6 weeks post-surgery
Population: Swab samples were able to be collected from all regions in all 9 patients in the Low-level therapy intervention arm and from all regions in all 8 patients in the Sham intervention arm who attended their Week 6 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 9 | 8
Participants
  R1 | 8 | 6
  R2 | 9 | 8
  R3 | 9 | 8
  R4 | 8 | 6
  L1 | 5 | 6
  L2 | 9 | 8
  L3 | 9 | 7
  L4 | 5 | 6

8. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 8 weeks post-surgery
Population: Swab samples were able to be collected from all regions in all 4 patients in the Low-level therapy intervention arm and from all regions in all 5 patients in the Sham intervention arm who attended their Week 8 visit. Due to a deviation one patient in the Sham group had swab samples collected at Week 7 instead of the intended 8-week timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 4 | 5
Participants
  R1 | 2 | 4
  R2 | 4 | 5
  R3 | 4 | 5
  R4 | 2 | 4
  L1 | 3 | 3
  L2 | 4 | 5
  L3 | 4 | 5
  L4 | 2 | 4

9. Primary Outcome: Inferior Alveolar Nerve Function for Soft Stimuli
Description: as for outcome 1
Time Frame: 20 weeks post-surgery
Population: Study was terminated in advance of the 20-week timepoint and swab samples were not collected from any of the participants at 20 weeks post-surgery. Accordingly, there are no IAN function for soft stimuli results to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: IAN function for hard stimuli was assessed by pressing a toothpick into the skin of the mandible and lower lip in 8 regions along the lower jaw. Regions right and left 1, 2, and 3 are on the skin of the lower face, 1 cm apart, starting on the midline, and right and left region 4 is the lower lip, separated at the midline. Right and left regions were abbreviated as R1, R2, R3, R4 and L1, L2, L3, and L4, respectively. Patients responded as to whether they were able to feel the toothpick using a binary Yes (+) or No (-) response. The number of patients who responded Yes (+) is summarized by study arm.
Time Frame: 24 hours post-surgery
Population: 24-hour post-surgical follow-up visits were not conducted during this study. Many patients were still admitted at 24 hours post-procedure and were unable to be brought into the dental clinic. In addition, the instruments and equipment required to conduct this assessment were not available in the hospital in-patient rooms. As a result, toothpick samples were not obtained from any of the patients at 24 hours post-surgery and there is no IAN function for hard stimuli results data to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 1 week post-surgery
Population: Toothpick samples were able to be collected from regions R1, R4, L1, and L4 in all 12 patients and from regions R2, R3, L2, and L3 in 11 of 12 patients in the Low-level therapy intervention arm who attended their Week 1 visit. Toothpick samples were able to be collected from regions R2, R3, L2, and L3 in all 8 patients and from regions R1, R4, L1, and L4 in 7 of 8 patients in the Sham intervention arm who attended their Week 1 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 12 | 8
Participants
  R1: number analyzed (Participants) | 12 | 7
  R1 | 10 | 2
  R2: number analyzed (Participants) | 11 | 8
  R2 | 11 | 8
  R3: number analyzed (Participants) | 11 | 8
  R3 | 11 | 8
  R4: number analyzed (Participants) | 12 | 7
  R4 | 7 | 2
  L1: number analyzed (Participants) | 12 | 7
  L1 | 8 | 0
  L2: number analyzed (Participants) | 11 | 8
  L2 | 11 | 6
  L3: number analyzed (Participants) | 11 | 8
  L3 | 11 | 8
  L4: number analyzed (Participants) | 12 | 7
  L4 | 8 | 4

12. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 2 weeks post-surgery
Population: Toothpick samples were able to be collected from all regions in all 10 patients in the Low-level therapy intervention arm who attended their Week 2 visit. Toothpick samples were able to be collected from all regions in all 9 patients in the Sham intervention arm with the exception of region L1 in which toothpick samples were able to be collected from 8 of 9 patients who attended their Week 2 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 10 | 9
Participants
  R1 | 6 | 5
  R2 | 10 | 9
  R3 | 10 | 9
  R4 | 7 | 5
  L1: number analyzed (Participants) | 10 | 8
  L1 | 6 | 5
  L2 | 10 | 8
  L3 | 10 | 9
  L4 | 5 | 5

13. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 3 weeks post-surgery
Population: Toothpick samples were able to be collected from all regions in all 10 patients in the Low-level therapy intervention arm and from all regions in all 8 patients in the Sham intervention arm who attended their Week 3 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 10 | 8
Participants
  R1 | 9 | 6
  R2 | 10 | 8
  R3 | 10 | 8
  R4 | 9 | 6
  L1 | 9 | 4
  L2 | 10 | 8
  L3 | 10 | 8
  L4 | 8 | 5

14. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 4 weeks post-surgery
Population: Toothpick samples were able to be collected from all regions in all 8 patients in the Low-level therapy intervention arm and from all regions in all 9 patients in the Sham intervention arm who attended their Week 4 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 8 | 9
Participants
  R1 | 5 | 7
  R2 | 8 | 9
  R3 | 8 | 9
  R4 | 7 | 8
  L1 | 4 | 6
  L2 | 8 | 9
  L3 | 8 | 9
  L4 | 5 | 5

15. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 5 weeks post-surgery
Population: Toothpick samples were able to be collected from regions L1 and L4 in all 7 patients and from regions R1, R2, R3, R4, L2, and L3 in 6 of 7 patients in the Low-level therapy intervention arm who attended their Week 5 visit. Toothpick samples were able to be collected from all regions in all 6 patients in the Sham intervention arm who attended their Week 5 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 7 | 6
Participants
  R1: number analyzed (Participants) | 6 | 6
  R1 | 6 | 3
  R2: number analyzed (Participants) | 6 | 6
  R2 | 6 | 6
  R3: number analyzed (Participants) | 6 | 6
  R3 | 6 | 6
  R4: number analyzed (Participants) | 6 | 6
  R4 | 5 | 3
  L1 | 3 | 4
  L2: number analyzed (Participants) | 6 | 6
  L2 | 6 | 6
  L3: number analyzed (Participants) | 6 | 6
  L3 | 6 | 6
  L4 | 3 | 3

16. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 6 weeks post-surgery
Population: Toothpick samples were able to be collected from all regions in all 9 patients in the Low-level therapy intervention arm and from all regions in all 8 patients in the Sham intervention arm who attended their Week 6 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 9 | 8
Participants
  R1 | 8 | 6
  R2 | 9 | 8
  R3 | 9 | 8
  R4 | 9 | 6
  L1 | 6 | 6
  L2 | 9 | 8
  L3 | 9 | 8
  L4 | 5 | 7

17. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 8 weeks post-surgery
Population: Toothpick samples were able to be collected from all regions in all 4 patients in the Low-level therapy intervention arm and from all regions in all 5 patients in the Sham intervention arm who attended their Week 8 visit. Due to a deviation one patient in the Sham group had toothpick samples collected at 7 weeks instead of the intended 8-week collection timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 4 | 5
Participants
  R1 | 2 | 4
  R2 | 4 | 5
  R3 | 4 | 5
  R4 | 2 | 4
  L1 | 3 | 4
  L2 | 4 | 5
  L3 | 4 | 5
  L4 | 2 | 4

18. Primary Outcome: Inferior Alveolar Nerve Function for Hard Stimuli
Description: as for outcome 10
Time Frame: 20 weeks post-surgery
Population: Study was terminated in advance of the 20-week timepoint and toothpick samples were not collected from any of the participants at 20 weeks post-surgery. Accordingly, there are no IAN function for hard stimuli results to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Post-operative Pain
Description: Post-operative pain was assessed and reported during each study visit using a single-item Visual Analog Scale (VAS) question. Patients rated the intensity of pain on each side of the mandible (right and left) on an 11-point Likert scale. Possible VAS scores ranged from 0 (complete absence of pain) to 10 (maximum amount of pain imaginable). Results were summarized by study arm using basic descriptive statistics.
Time Frame: 24 hours post-surgery
Population: 24-hour post-surgical follow-up visits were not conducted during this study. Many patients were still admitted at 24 hours post-procedure and were unable to be brought into the dental clinic. In addition, the instruments and equipment required to conduct this assessment were not available in the hospital in-patient rooms. As a result, VAS scores were not obtained from any of the patients at 24 hours post-surgery and there are no post-operative pain results data to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 1 week post-surgery
Population: 1-week post-operative pain (VAS) data was able to be collected from all 12 patients in the Low-level therapy intervention arm and from all 8 patients in the Sham intervention arm who attended their Week 1 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 12 | 8
score on a scale
  Right Side | 2.6 (2.2) | 2.3 (3.1)
  Left Side | 1.9 (1.9) | 1.0 (1.7)

21. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 2 weeks post-surgery
Population: 2-week post-operative pain (VAS) data was able to be collected from 9 of 10 patients in the Low-level therapy intervention arm and from all 9 patients in the Sham intervention arm who attended their Week 2 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 9 | 9
score on a scale
  Right Side | 1.1 (1.3) | 1.4 (2.2)
  Left Side | 1.4 (2.2) | 0.8 (1.1)

22. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 3 weeks post-surgery
Population: 3-week post-operative pain (VAS) data was able to be collected from 9 of 10 patients in the Low-level therapy intervention arm and from all 8 patients in the Sham intervention arm who attended their Week 3 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 9 | 8
score on a scale
  Right Side | 0.9 (0.8) | 1.5 (1.8)
  Left Side | 1.3 (1.7) | 1.3 (1.7)

23. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 4 weeks post-surgery
Population: 4-week post-operative pain (VAS) data was able to be collected from all 8 patients in the Low-level therapy intervention arm and from all 9 patients in the Sham intervention arm who attended their Week 4 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 8 | 9
score on a scale
  Right Side | 1.0 (1.3) | 0.3 (0.5)
  Left Side | 0.5 (0.5) | 0.3 (0.5)

24. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 5 weeks post-surgery
Population: 5-week post-operative pain (VAS) data was able to be collected from all 7 patients in the Low-level therapy intervention arm and from all 6 patients in the Sham intervention arm who attended their Week 5 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 7 | 6
score on a scale
  Right Side | 0.7 (0.8) | 0.8 (1.2)
  Left Side | 0.6 (0.5) | 0.8 (1.2)

25. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 6 weeks post-surgery
Population: 6-week post-operative pain (VAS) data was able to be collected from all 9 patients in the Low-level therapy intervention arm and from all 8 patients in the Sham intervention arm who attended their Week 6 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 9 | 8
score on a scale
  Right Side | 0.3 (0.5) | 0.5 (0.5)
  Left Side | 0.3 (0.5) | 0.4 (0.5)

26. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 8 weeks post-surgery
Population: 8-week post-operative pain (VAS) data was able to be collected from all 4 patients in the Low-level therapy intervention arm and from all 5 patients in the Sham intervention arm who attended their Week 8 visit. Due to a deviation one patient in the Sham group had VAS data collected at 7 weeks instead of the intended 8-week collection timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 4 | 5
score on a scale
  Right Side | 0.5 (0.6) | 0.2 (0.4)
  Left Side | 0.5 (0.6) | 0.2 (0.4)

27. Secondary Outcome: Post-operative Pain
Description: as for outcome 19
Time Frame: 20 weeks post-surgery
Population: Study was terminated in advance of the 20-week timepoint and the VAS questionnaire was not administered to, nor were data collected from, any of the participants at 20 weeks post-surgery. Accordingly, there are no post-operative pain results to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Post-operative Mandibular Swelling
Description: Post-operative mandibular swelling was measured using soft measuring tape. The extent of post-operative swelling was measured from the tip of the chin to the base of the earlobe bilaterally (right and left). Measurements were recorded in millimeters (mm) and results summarized by study arm using basic descriptive statistics.
Time Frame: 24 hours post-surgery
Population: 24-hour post-surgical follow-up visits were not conducted during this study. Many patients were still admitted at 24 hours post-procedure and were unable to be brought into the dental clinic. In addition, the instruments and equipment required to conduct this assessment were not available in the hospital in-patient rooms. As a result, mandibular swelling measurements were not obtained from any of the patients at 24 hours post-surgery and there is no mandibular swelling results data to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 1 week post-surgery
Population: 1-week post-operative mandibular swelling data was able to be collected from all 12 patients in the Low-level therapy intervention arm and from all 8 patients in the Sham intervention arm who attended their Week 1 visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 12 | 8
millimeters
  Right Side | 153 (12.3) | 138 (23.7)
  Left Side | 156 (16.4) | 133 (25.7)

30. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 2 weeks post-surgery
Population: 2-week post-operative mandibular swelling data was able to be collected from all 10 patients in the Low-level therapy intervention arm and from all 9 patients in the Sham intervention arm who attended their Week 2 visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 10 | 9
millimeters
  Right Side | 154 (18.0) | 140 (18.8)
  Left Side | 152 (23.0) | 132 (27.3)

31. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 3 weeks post-surgery
Population: 3-week post-operative mandibular swelling data was able to be collected from all 10 patients in the Low-level therapy intervention arm and from 7 of 8 patients in the Sham intervention arm who attended their 3-week visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 10 | 7
millimeters
  Right Side | 145 (12.7) | 134 (21.3)
  Left Side | 142 (13.8) | 135 (21.8)

32. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 4 weeks post-surgery
Population: 4-week post-operative mandibular swelling data was able to be collected from all 8 patients in the Low-level therapy intervention arm and from all 9 patients in the Sham intervention arm who attended their Week 4 visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 8 | 9
millimeters
  Right Side | 147 (7.41) | 146 (12.2)
  Left Side | 149 (10.5) | 142 (16.9)

33. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 5 weeks post-surgery
Population: 5-week post-operative mandibular swelling data was able to be collected from all 7 patients in the Low-level therapy intervention arm and from all 6 patients in the Sham intervention arm who attended their Week 5 visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 7 | 6
millimeters
  Right Side | 152 (13.1) | 134 (32.0)
  Left Side | 151 (16.0) | 134 (31.1)

34. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 6 weeks post-surgery
Population: 6-week post-operative mandibular swelling data was able to be collected from all 9 patients in the Low-level therapy intervention arm and from all 8 patients in the Sham intervention arm who attended their Week 6 visit.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 9 | 8
millimeters
  Right Side | 145 (15.2) | 141 (15.0)
  Left Side | 141 (15.8) | 139 (16.7)

35. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 8 weeks post-surgery
Population: 8-week post-operative mandibular swelling data was able to be collected from all 4 patients in the Low-level therapy intervention arm and from all 5 patients in the Sham intervention arm who attended their Week 8 visit. Due to a deviation one patient in the Sham group had Post-operative mandibular swelling data collected at 7 weeks instead of the intended 8-week collection timepoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 4 | 5
millimeters
  Right Side | 139 (10.8) | 136 (19.2)
  Left Side | 134 (14.8) | 135 (21.3)

36. Secondary Outcome: Post-operative Mandibular Swelling
Description: as for outcome 28
Time Frame: 20 weeks post-surgery
Population: Study was terminated in advance of the 20-week timepoint and post-operative mandibular swelling measurements were not collected from any of the participants at 20 weeks post-surgery. Accordingly, there are no post-operative mandibular swelling results to report.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 8 weeks post-surgical intervention.
Arm/Group | Low-level Therapy Intervention | Sham Intervention
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT04910074/Prot_SAP_002.pdf